CLINICAL TRIAL: NCT06428318
Title: Diagnostic Value of the Biofire® Filmarray Pneumonia Panel Compared to Conventional Sputum Culture in Critically il Patients With Pneumonia
Brief Title: Diagnostic Value of the Biofire®in Community Acquired Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rania Maher Hussien, MD, Associate Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: FMASU MS267/2023
Record Dates: First submitted 2024-05-21; First posted 2024-05-24 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Routine Conventional Methods (Active Comparator): Patients subjected to Routine sputum culture Conventional Methods
  Interventions: Diagnostic Test: Conventional Sputum culture
- GroupB: BioFire Pneumonia Panel (BFPP). (Active Comparator): Patients subjected to BioFire Pneumonia Panel (BFPP
  Interventions: Diagnostic Test: BioFire Pneumonia Panel (BFPP)

INTERVENTIONS:
Diagnostic Test: Conventional Sputum culture — Sputum culture was done to patients and they received Antibiotics According to its results
  Arms: Group A: Routine Conventional Methods
Diagnostic Test: BioFire Pneumonia Panel (BFPP) — BioFire Pneumonia Panel (BFPP) was done to patients and they received Antibiotics According to its results
  Arms: GroupB: BioFire Pneumonia Panel (BFPP).

SUMMARY:
This study aimed to determine the impact value of the BioFire FilmArray Pneumonia panel compared to conventional sputum culture in critically ill patients with pneumonia.

DETAILED DESCRIPTION:
the BioFire® FilmArray Pneumonia Panel (BFPP) emerges as a promising candidate for a rapid and multifaceted diagnostic approach.

This study compare the diagnostic accuracy, turnaround time, and impact on antibiotic management decisions of BFPP versus conventional sputum culture in critically ill patients admitted to the ICU with suspected pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the ICU with community acquired pneumonia

Exclusion Criteria:

* Age less than 18 years old.
* End stage malignant patients,
* Patients admitted to the ICU with Acute Lung Injury (ALI).
* Patients admitted to the ICU with Acute Respiratory Distress Syndrome (ARDS).
* Patients with radiological findings suggesting atypical pneumonia.
* Immunocompromised as defined by HIV/AIDS, known immunodeficiency, chronic steroids > 20mg/day Prednisone equivalent, other immunosuppressants.
* Solid organ or bone marrow transplant patients, cystic fibrosis.
* Unstable psychiatric or psychological condition rendering the subject unlikely to be cooperative or to complete the study requirements.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
the ICU length of stay | Five days after admission
  The potential correlation between the use of BFPP and its relation to the ICU length of stay

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Abassia, Egypt